CLINICAL TRIAL: NCT03642795
Title: Validation of the French Version of the CQR (Compliance Questionnaire Rheumatology): Specific Tool for Evaluation of Observance of Rheumatology Treatment
Brief Title: Validation of the French Version of the CQR (Compliance Questionnaire Rheumatology)
Acronym: CQR-F
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRCI/2016/CGV-01
Record Dates: First submitted 2017-11-14; First posted 2018-08-22 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Polyarthritis
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with rheumatoid polyarthritis
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients are asked to complete several questionnaires

SUMMARY:
The purpose of this study is to develop a French language version of the Compliance-Questionnaire-Rheumatology for use in French and Francophone rheumatology services

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* The patient is at least 18 years old
* The patient has rheumatoid polyarthritis as defined by the ACR-EULAR 2010 criteria, treated orally or subcutaneously with MTX for at least 3 months with a stable (unchanged) dosage for at least 1 month, and a stable (unchanged) route of administration for at least 1 month. And no planned change in Methotrexate intake at least until the second study visit. Other treatments at the same time are authorized

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The subject has a contraindication to taking methotrexate (including a patient with a desire to become pregnant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid polyarthritis as defined by the ACR-EULAR 2010 criteria, treated orally or subcutaneously with MTX for at least 3 months being followed in the rheumatology department of Montpellier, Toulouse, Bordeaux or Nîmes hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Test-retest agreement of French translation of the Compliance Questionnaire Rheumatology questionnaire | 40 minutes
  Intraclass correlation and Kappa coefficient of 2 evaluations taken 40 minutes apart
Structural validity of French translation of the Compliance Questionnaire Rheumatology questionnaire | Baseline
  Principal component analysis

SECONDARY OUTCOMES:
Validation of the Compliance Questionnaire Rheumatology against gold standard (erythrocyte methotrexate polyglutamates (MTX PGs) concentration) | Baseline
  CQR ≥80% (observant) vs MTX PGs level
Rate of missing responses to each question of French translation of Compliance Questionnaire Rheumatology | Baseline
  %
Rate of questionnaires with at least 1 missing item | Baseline
  %
Validation of the short form of the French Compliance Questionnaire Rheumatology | Baseline
  5-item questionnaire
Compare French Compliance Questionnaire Rheumatology results against general questionnaire Morisky Medication Adherence Scale (MMAS-8) | Baseline
  Sensitivity and specificity compared against MTX PGs level
Sex of observant versus non-observant patients | Month 1
  male/female
Age of observant versus non-observant patients | Month 1
  years
education level of observant versus non-observant patients | Month 1
  school graduation
profession of observant versus non-observant patients | Month 1
  name of the profession
marital status of observant versus non-observant patients | Month 1
  Married, single, divorced, widowed
Number patients observing medication | Month 1
  Blood MTX PG concentration nmol/L by LC-MS/MS
Quality of life in observant versus non-observant patients | Month 1
  Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
Health-related quality of life in observant versus non-observant patients | Month 1
  Euroqol 5 dimension 3 level questionnaire (EQ5D-3L)
Functional incapacity in observant versus non-observant patients | Month 1
  Health Assessment Questionnaire (HAQ)
Pain experience in observant versus non-observant patients | Month 1
  Pain Catastrophizing Scale (PCS-CF)
Cognitive representations of medication in observant versus non-observant patients | Month 1
  Beliefs about Medicines Questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU Bordeaux, Bordeaux
  - CHRU Montpellier, Montpellier
  - CHU Nimes, Nîmes
  - CHU Toulouse, Toulouse